CLINICAL TRIAL: NCT01128829
Title: Regulation of Incretin Release by Non-nutritive Sweeteners in Humans
Brief Title: Sugar-replacement Sweeteners, and Blood Sugar Control
Acronym: SIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Marta Yanina Pepino de Gruev, Research Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0583/ 201102383
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
Keywords: obesity; diabetes; artificial sweeteners
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Water; trichlorosucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water-sucralose (Experimental): Subjects in this group drank "water" 10 min before drinking a glucose load on their first oral glucose tolerance test (OGTT) and drank "sucralose" 10 min before drinking a glucose load on their second OGTT. The two OGTT were separated on average by 1 week (i.e. washout was approximately 1 week).
  Interventions: Other: Water; Other: Sucralose
- sucralose-water (Experimental): Subjects in this group drank "sucralose" 10 min before drinking a glucose load on their first OGTT and drank "water" 10 min before drinking a glucose load on their second OGTT. The two OGTT were separated on average by 1 week (i.e. washout was approximately 1 week).
  Interventions: Other: Water; Other: Sucralose

INTERVENTIONS:
Other: Water — 60 ml of water were drank 10 min before doing a OGTT
Other: Sucralose — 60 ml of 2 millimolar sucralose were drank 10 min before doing a OGTT

SUMMARY:
Several sugar-replacement sweeteners are currently on the market, including saccharine (ex. Sweet'N Low), aspartame (ex. Equal), and sucralose (ex. Splenda). The purpose of this study is to examine wether non caloric sweeteners affects how well the body works to control blood sugar. The study includes detailed blood sugar testing after drinking liquids that may contain sucralose. The investigators hypothesize that drinking liquids with sucralose will effect the amounts of specific appetite-affecting substances naturally produced by the body.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) over 30.
* Homeostasis model assessment of insulin resistance (HOMA-IR) < or = 2.6

Exclusion Criteria:

* smoking or smoked within last six months
* pregnant or breastfeeding
* have malabsorptive syndromes
* intestinal inflammatory disease
* diabetes
* liver or kidney disease
* fructose intolerance
* consuming more than one can of diet beverage or one spoonful of non-nutritive sweeteners (e.g. sucralose, aspartame, or saccharine) a week.
* taking any medication that might affect metabolism or taste.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-05; Primary Completion 2012-02 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Y Pepino de Gruev, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Pepino MY, Tiemann CD, Patterson BW, Wice BM, Klein S. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes Care. 2013 Sep;36(9):2530-5. doi: 10.2337/dc12-2221. Epub 2013 Apr 30. PMID 23633524

RESULTS

PARTICIPANT FLOW:
Groups:
- "Water Then Sucralose": First intervention (1 day) subjects drank 60 ml of water 10 min before drinking a 75 g glucose load.
  Washout (~ 7 days) Second intervention (1 day) subjects drank 60 ml of 2 mmolar sucralose 10 min before drinking a 75 g glucose load.
- "Sucralose Then Water": First intervention (1 day) subjects drank 60 ml of 2 mmolar sucralose10 min before drinking a 75 g glucose load.
  Washout (~ 7 days) Second intervention (1 day) subjects drank 60 ml of water 10 min before drinking a 75 g glucose load.
Period: Overall Study
Arm/Group | "Water Then Sucralose" | "Sucralose Then Water"
Started | 6 | 11
Completed | 6 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Obese Non Regular Users of Non Nutritive Sweeteners (NNS): Obese subjects who do not use NNS and are "insulin-sensitive" (based on a Homeostasis Model Assessment of Insulin Resistance score <or =2.6).
Arm/Group | Obese Non Regular Users of Non Nutritive Sweeteners (NNS)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Sucralose on Insulin Concentration (Area Under the Curve; AUC)
Description: we will measure plasma insulin concentrations during a 5-hour modified Oral Glucose Tolerance Test (mOGTT) administered 10 minutes after subjects consume sucralose in water or an equal volume of water without sucralose (control condition).Plasma insulin concentrations were measured at 20, 15, 10, 6, and 2 min before and at 10, 20, 30, 40, 60, 90, 120, 150,180, 240, and 300 min after ingesting 75g of glucose. All these data collected were used to create the AUC curve.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: (pmol • min •L-1)
Arm/Group | Obese Non Regular Users of Non Nutritive Sweeteners (NNS)
Number analyzed (Participants) | 17
(pmol • min •L-1)
  Insulin AUC on water day | 57,192 (23,270)
  Insulin AUC on sucralose day | 68,647 (31,201)
Statistical Analysis 1: Comparison: Obese Non Regular Users of Non Nutritive Sweeteners (NNS); Each subject served as their own control. We compared insulin concentrations when subjects consumed sucralose before a glucose load (experimental condition) with those on the day consumed water before a glucose load (control condition); Test type: Superiority or Other; p = 0.025, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Obese Non Regular Users of Non Nutritive Sweeteners (NNS)
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No